CLINICAL TRIAL: NCT04868656
Title: Implementing a Hospital-Based Walking Program (STRIDE): Function QUERI 2.0 (QUE 20-023)
Brief Title: Implementing a Hospital-Based Walking Program (STRIDE): Function QUERI 2.0
Acronym: STRIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: QUX 21-001
Record Dates: First submitted 2021-04-27; First posted 2021-05-03 (Actual); Results first posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Early Ambulation
Keywords: Walking; Veterans; Inpatients; Quality of Life; Implementation Science; Functional Independence; Early Ambulation

STUDY DESIGN:
Intervention Model Description: Parallel cluster-randomized trial (parallel-CRT): used in pragmatic evaluations of health program or policy interventions, where half the clusters (in this case, VA hospitals) are randomly assigned to two interventions: Foundational support (active comparator) vs. Enhanced support (experimental).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Foundational Support (Active Comparator): Foundational Support uses the Replicating Effective Program (REP) implementation strategy and includes 5 elements that were developed and tested in our prior Function QUERI work: STRIDE Toolkit; Online shared resources (SharePoint) access for clinical program training materials; Data dashboard to assist hospitals with tracking their own data; Diffusion Networks to promote peer-to-peer sharing and implementation support; and Microsoft TEAMS Channels.
  Interventions: Other: Implementation Strategy: Foundational Support
- Enhanced Support (Experimental): Enhanced Support begins with the same activities as Foundational Support. Hospitals that are randomized to Enhanced Support and do not meet STRIDE initial program benchmarks within 6 months will continue with Foundational support and also receive higher intensity support for a period of 4-6 months. Hospitals that have sustained their implementation will continue low-touch activities while those that have been randomized to the enhanced support arm and met the initial program benchmark at 6-months but have not sustained (did not meet the sustainment benchmark), will begin engaging in high-touch activities. The higher intensity support will consist of facilitation, a process of interactive problem solving and support that occurs in a context of a supportive interpersonal relationship. Facilitation will be provided by Function QUERI team members.
  Interventions: Other: Implementation Strategy: Enhanced Support

INTERVENTIONS:
Other: Implementation Strategy: Foundational Support — The goal is to test implementation intensification approaches for STRIDE hospitals that have not met implementation program benchmarks, specifically Foundational Support vs. Enhanced Support. We propose that low intensity implementation support that promotes adapting STRIDE for context and provides tools for ongoing STRIDE evaluation (defined as foundational support), will be sufficient for some but not all hospitals to successfully incorporate STRIDE into routine practice.
  Other Names: Foundational REP
  Arms: Foundational Support
Other: Implementation Strategy: Enhanced Support — The goal is to test implementation intensification approaches for STRIDE hospitals that have not met implementation program benchmarks, specifically Foundational Support vs. Enhanced Support. We posit that monitoring hospitals' progress and adding, for hospitals with low adoption, higher intensity strategies (defined as Enhanced Support) that directly influence teams' capacity and skills to effectively self-organize and problem-solve will lead to higher implementation adoption, penetration, fidelity, and value.
  Other Names: Enhanced REP
  Arms: Enhanced Support

SUMMARY:
Implementing a Hospital-Based Walking Program (STRIDE): Function QUERI 2.0 aims to compare implementation strategies for large-scale spread of STRIDE, a supervised walking program for hospitalized older Veterans. The overall goal is to implement, evaluate, and sustain STRIDE in 32 additional VA hospitals using a type III effectiveness-implementation hybrid design framework.

DETAILED DESCRIPTION:
Background/Purpose. Hospitalization is a major risk factor for development of disability. More than one-third of adults over the age of 70 are discharged from the hospital with a major new disability that was not present before the onset of acute illness. A key contributor to hospital-associated disability is immobility during hospitalization. Although fewer than 5% of patients have physician orders for bed rest, hospitalized older adults spend only about 3% of their time standing or walking. The hazards of bedrest have been recognized for more than 2 decades, but there remains a persistent 'epidemic of immobility' in American hospitals.

STRIDE is a supervised inpatient walking program developed by an interdisciplinary team of investigators, clinicians and administrators at the Durham VA and funded by the Veterans Health Administration (VHA) Office of Geriatrics and Extended Care. STRIDE is designed for patients aged >= 60 years and consists of a one-time gait and balance assessment, followed by daily walks supervised by a mobility assistant for the duration of the hospital stay. Clinical demonstration of STRIDE conducted at the Durham VA resulted in a greater likelihood of discharge to home than to skilled nursing or rehabilitation among STRIDE participants compared to clinically similar patients receiving usual care. Based on this experience, the cumulative evidence of the positive impact of early mobility interventions, and successful spread to other hospitals, STRIDE has the potential to become a system-wide approach to address hospital-associated disability in VA.

As part of Implementing a Hospital-Based Walking Program (STRIDE), the investigators plan to implement the STRIDE clinical program at an additional 32 VA hospitals using a type III effectiveness-implementation hybrid design framework with hospitals enrolled and randomized to receive low-touch implementation support (foundational support) or a higher-intensity implementation support (enhanced support including additional facilitation, self-organization, and team building support) for hospitals that do not meet program benchmarks at 6 and 8 months.

Objectives. The investigators plan to develop scalable approaches to implement and sustain STRIDE as well as evaluate implementation with foundational support versus the enhanced-implementation strategy (enhanced support).

Key questions: How should the STRIDE clinical program be adapted to optimize sustainability? Are there differences in implementation outcomes (penetration, fidelity) at 10 months (primary), 13, 16 months between arms? How do hospitals experience implementation strategies in each arm? What baseline organizational characteristics are associated with hospitals that do not meet implementation benchmarks? The investigators also plan to conduct an explanatory sequential mixed method design that includes qualitative data collection and analysis that will not be reported here. Additionally, adoption will be examined at 10 months.

Methodology. To evaluate implementation, the investigators will randomize hospitals (n=32) 1:1 to either foundational support or enhanced support. The investigators will use generalized linear models to examine the effect of foundational vs. enhanced on implementation outcomes at 10-months.

ELIGIBILITY:
Inclusion Criteria:

* Hospital inclusion criteria includes submission of a signed participation agreement.

  * All enrolled hospitals will all be exposed to Foundational Support.
  * Hospitals randomized to Enhanced Support that do not meeting STRIDE initial program benchmarks will receive higher-intensity implementation support (Enhanced Support).
* The clinical outcomes assessment will include all patients >=60 that have an admission on a general medicine ward that offers STRIDE program at enrolled site.

Exclusion Criteria:

* The eight STRIDE hospitals that have previously participated in Function QUERI (ClinicalTrials.gov Identifier: NCT03300336) will be excluded from enrollment in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan N. Hastings, MD MHSc, Principal Investigator — Durham VA Medical Center, Durham, NC; Courtney H Van Houtven, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC; Kelli Dominick Allen, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be available upon request. Prior to distribution, a local privacy officer and study statistician will certify that the dataset contains no protected health information (PHI). Data will be provided to requestor in electronic format. Sufficient data and descriptors will be made available to duplicate statistical analysis and confirm conclusions in publication. No data or statistical code that could lead to re-identification of individuals will be released. Data will be stored & maintained in an approved, secured location as described in the VA Research Data Inventory Form. The statistician will create de-identified, publication-specific datasets that includes variables from statistical models presented in publication. Data will only be released per appropriate authorizations or agreements. Written agreements will specify that recipients are prohibited from taking steps to re-identify any individual whose data are included in the dataset.
Supporting Information: Study Protocol
Time Frame: Available upon request.
Access Criteria: Data will only be released per appropriate authorizations or agreements. Written agreements will specify that recipients are prohibited from taking steps to re- identify any individual whose data are included in the dataset.

REFERENCES:
- [Derived] Kappler CB, Coffman CJ, Stechuchak KM, Choate A, Meyer C, Zullig LL, Hughes JM, Drake C, Sperber NR, Kaufman BG, Van Houtven CH, Allen KD, Hastings SN. Evaluation of strategies to support implementation of a hospital walking program: protocol for a type III effectiveness-implementation hybrid trial. Implement Sci Commun. 2024 Jan 12;5(1):8. doi: 10.1186/s43058-024-00544-5. PMID 38216967
- [Derived] Hughes JM, Zullig LL, Choate AL, Decosimo KP, Wang V, Van Houtven CH, Allen KD, Nicole Hastings S. Intensification of Implementation Strategies: Developing a Model of Foundational and Enhanced Implementation Approaches to Support National Adoption and Scale-up. Gerontologist. 2023 Mar 21;63(3):604-613. doi: 10.1093/geront/gnac130. PMID 36029028

RESULTS

PARTICIPANT FLOW:
Recruitment Details: VA hospitals were enrolled in five successive cohorts from June 1, 2021 to October 3, 2022.
Units Other Than Participants: Hospital
Period: Overall Study
Arm/Group | Foundational Support | Enhanced Support
Started | NA; 19 Hospital (Data was collected at the VA site level) | NA; 16 Hospital (Data was collected at the VA site level)
Completed | NA; 19 Hospital (Data was collected at the VA site level) | NA; 16 Hospital (Data was collected at the VA site level)
Not Completed | NA; 0 Hospital | NA; 0 Hospital

BASELINE CHARACTERISTICS:
Population: Data was collected at the site level and these characteristics were not relevant and not collected.
Units Other Than Participants: Hospital
Groups:
- Total: Total of all reporting groups
Arm/Group | Foundational Support | Enhanced Support | Total
Number analyzed (Participants) | NA | NA | NA
Number analyzed (Hospital) | 19 | 16 | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Data was collected at the site level and these characteristics were not relevant and not collected.
  Years
    number analyzed (Hospital) | 0 | 0 | 0
Sex: Female, Male [Count of Units; unit: Hospital] — Population: Data was collected at the site level and these characteristics were not relevant and not collected.
  Hospital
    number analyzed (Hospital) | 0 | 0 | 0
    Female |  |  | 0
    Male |  |  | 0
Race (NIH/OMB) [Count of Units; unit: Hospital]
  American Indian or Alaska Native | NA — Data was collected at the site level and these characteristics were not relevant and not collected. | NA — Data was collected at the site level and these characteristics were not relevant and not collected. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Asian | NA — Data was collected at the site level and these characteristics were not relevant and not collected. | NA — Data was collected at the site level and these characteristics were not relevant and not collected. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Native Hawaiian or Other Pacific Islander | NA — Data was collected at the site level and these characteristics were not relevant and not collected. | NA — Data was collected at the site level and these characteristics were not relevant and not collected. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black or African American | NA — Data was collected at the site level and these characteristics were not relevant and not collected. | NA — Data was collected at the site level and these characteristics were not relevant and not collected. | NA — Total not calculated because data are not available (NA) in one or more arms.
  White | NA — Data was collected at the site level and these characteristics were not relevant and not collected. | NA — Data was collected at the site level and these characteristics were not relevant and not collected. | NA — Total not calculated because data are not available (NA) in one or more arms.
  More than one race | NA — Data was collected at the site level and these characteristics were not relevant and not collected. | NA — Data was collected at the site level and these characteristics were not relevant and not collected. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | NA — Data was collected at the site level and these characteristics were not relevant and not collected. | NA — Data was collected at the site level and these characteristics were not relevant and not collected. | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: Hospital]
  United States : Northeast | 3 | 3 | 6
  United States : Midwest | 5 | 5 | 10
  United States : South | 5 | 3 | 8
  United States : West | 6 | 5 | 11
Facility Complexity Scores [Count of Units; unit: Hospital] — 1a is the most complex versus all others.
  Hospital
    1a | 8 | 6 | 14
    1b, 1c, 2 , 3 | 11 | 10 | 21
Adjusted Length of Stay [Count of Units; unit: Hospital]
  Greater than or equal to 4.7 days | 12 | 10 | 22
  Less than 4.7 days | 7 | 6 | 13
Prior Mobility Program Experience [Count of Units; unit: Hospital]
  Yes | 6 | 5 | 11
  No | 13 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: Penetration
Description: Penetration is defined as the percent of eligible hospitalizations with one or more STRIDE walks at 10 months. It is not possible to assess all eligibility criteria in the Electronic Health Record (e.g. able to walk at baseline); thus, with this more inclusive denominator, 100% penetration is not an appropriate goal. Based on preliminary data, we anticipate penetration to range from 0% (no program activity at 10-month outcome assessment) to 40% (estimated maximum achievable based on data from current STRIDE sites).
Time Frame: 10 months (cumulative)
Population: Data collected at the site level
Measure: Mean (Standard Deviation); unit: percentage of eligible hospitalizations
Units Other Than Participants: Hospital
Arm/Group | Foundational Support | Enhanced Support
Number analyzed (Participants) | NA | NA
Number analyzed (Hospital) | 19 | 16
percentage of eligible hospitalizations | 4.3 (4.7) | 2.2 (3.0)
Statistical Analysis 1: Comparison: Foundational Support vs Enhanced Support; Models included the arm indicator variable in addition to the stratification variables used in randomization (site complexity level (high complexity '1a', '1b' or '1c' vs. all others); adjusted length of stay (greater than or equal to 4.7 days versus less than 4.7 days); prior implementation of STRIDE (yes vs. no); Test type: Superiority; p = 0.15, Regression, Linear; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-5.0 to 0.8]

2. Secondary Outcome: Fidelity
Description: Fidelity will be the percentage of eligible hospital days with "full dose" of the program, defined as two or more documented walks or one walk for more than five minutes.
Time Frame: 10 months (cumulative)
Population: Data collected at the site level
Measure: Mean (Standard Deviation); unit: percentage of eligible hospital days
Units Other Than Participants: Hospital
Arm/Group | Foundational Support | Enhanced Support
Number analyzed (Participants) | NA | NA
Number analyzed (Hospital) | 19 | 16
percentage of eligible hospital days | 35 (10) | 40 (14)
Statistical Analysis 1: Comparison: Foundational Support vs Enhanced Support; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.34, Regression, Linear; Mean Difference (Final Values) = 5.3, 95% CI 2-sided [-6.0 to 16.6]

3. Secondary Outcome: Adoption
Description: Program adoption is a binary outcome defined for each hospital as equal to or more than 5 patients with a STRIDE walk or not.
Time Frame: 10 months (cumulative)
Population: Data collected at the site level
Measure: Number; unit: Hospitals with Program Adoption
Units Other Than Participants: Hospitals
Arm/Group | Foundational Support | Enhanced Support
Number analyzed (Participants) | NA | NA
Number analyzed (Hospitals) | 19 | 16
Hospitals with Program Adoption | 13 | 9
Statistical Analysis 1: Comparison: Foundational Support vs Enhanced Support; Model includes the arm indicator variable only; model does not include stratification variables due to potential for overfitting; Test type: Superiority; p = 0.23, Regression, Logistic; Odds Ratio (OR) = 0.6, 95% CI 2-sided [0.1 to 2.5]

ADVERSE EVENTS:
Time Frame: Analysis was at the site level and there were no possible adverse events.
Description: All cause mortality and/or serious adverse or other (Not Including Serious) adverse events were not collected on Veterans, caregivers, or providers.
Arm/Group | Foundational Support | Enhanced Support
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT04868656/Prot_SAP_001.pdf
  • Informed Consent Form (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/56/NCT04868656/ICF_000.pdf